CLINICAL TRIAL: NCT04914377
Title: A Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety and Efficacy of TQ Formula in Treating Participants Who Have Tested Positive for Novel Coronavirus 2019 (BOSS-Covid-19)
Brief Title: To Evaluate the Safety and Efficacy of TQ Formula in Covid-19 Participants
Acronym: BOSS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novatek Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BOSS-001
Record Dates: First submitted 2021-06-02; First posted 2021-06-04 (Actual); Results first posted 2024-08-14 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-07

CONDITIONS: Covid19
Keywords: TQ Formula; Covid 19
MeSH Terms: conditions — COVID-19 | interventions — Nigella sativa oil

STUDY DESIGN:
Intervention Model Description: This is a randomized, double-blind, placebo-controlled phase II study to assess the safety and efficacy of TQ Formula versus placebo in the treatment of Covid-19 in an outpatient setting. Participants will be randomized 1:1 to receive either 3 g per day of TQ Formula or placebo (identical in appearance). The participants will receive up to 14 days of dosing.
Who Masked: Participant, Investigator
Masking Description: Double-blind study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Active Drug (Experimental): Capsules containing TQ Formula
  Interventions: Drug: TQ Formula/Tab
- Placebo (Placebo Comparator): Capsules containing corn oil
  Interventions: Drug: TQ Formula/Tab

INTERVENTIONS:
Drug: TQ Formula/Tab — TQ Formula will be administered as an oral dose daily. The dose planned in this study is 3 g per day (3 500mg capsules to be taken twice daily).
  Other Names: Nigella Sativa

SUMMARY:
This is a randomized (1:1), double-blind, placebo-controlled phase 2 study to assess safety and efficacy of Total TQ Formula (3 g daily dose of Nigella Sativa Oil) capsules versus placebo in treating patients who have tested positive for novel Coronavirus 2019 (Covid-19) in the outpatient setting.

Patients will be treated at a dose of 500 mg, 3 capsules, two times a day for 14 days from date of randomization. Quantitative viral load as measured by RT-PCR will be evaluated at baseline and on days 7 and 14. Covid-19 symptoms will be measured throughout the study using Modified FLU-PRO Plus.

DETAILED DESCRIPTION:
Study Population: Up to 60 participants will be randomized 1:1 to receive either TQ Formula Capsules + Standard of Care (SOC) or placebo +SOC

Phase: Phase II

Approximately 2-4 centers in the United States

TQ Formula (Nigella Sativa) 500 mg, 3 capsules, BID, taken orally

Study Duration: 6 months

Participant Duration: Up to 45 days

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Male or female, aged 18 and over, presenting with recent mild to moderate clinical symptoms of Covid-19 infection (per FDA guidance - see appendix 3)
4. Positive COVID-19 infection confirmed with a rapid antigen test at screening (or RT-PCR within the last 3 days) and confirmed with a RT-PCR test at baseline
5. A score of >/=3 on a minimum of 2 symptoms on the Modified FLU-PRO Plus
6. Ability to take oral medication and be willing to adhere to the dosing regimen (Twice a day - BID for 14 days)
7. For females of reproductive potential: negative pregnancy test at screening and use of highly effective contraception method during study participation and for an additional 4 weeks after the end of study drug administration
8. For males of reproductive potential: use of condoms or other methods to ensure effective contraception with partner during study participation
9. Agreement to adhere to Lifestyle Considerations (see section 5.3) throughout study duration

Exclusion Criteria:

1. Current or recent (within 4 weeks) treatment with any corticosteroids; however, high-dose inhaled steroids, which are used to treat acute or chronic bronchial inflammation, will be permitted
2. Current or recent (within 4 weeks) treatment with any antivirals
3. Room air oxygen saturation (SaO2) < 94% at screen
4. Walking oximetry < 90% or participant unable to complete 6-minute walking oximetry test at screen
5. Severe Covid-19 symptoms (severe per FDA classification - see appendix 3)
6. Requires immediate admission to hospital for any reason
7. Pregnancy or lactation
8. Known allergic reactions to components of black seed oil, or thymoquinone
9. Treatment with another investigational drug or other investigational intervention within 2 weeks of study start and throughout study duration.
10. Significant hepatic disease (ALT/AST> 4 times the ULN); any laboratory parameter >/= 4 times the ULN
11. History of moderate to severe CKD, (i.e. an estimated glomerular filtration rate less than 45 mL/min) at the time of enrollment or history of liver disease
12. Patients with inflammatory bowel disease (such as Crohn's) that could affect the intestinal absorption of TQ Formula enteric coated capsules.
13. Known HIV or Hepatitis C infection
14. Influenza diagnosis (confirmed by testing) during screening or within prior 14 days
15. Any uncontrolled condition(s) or diagnosis, both physical or psychological, or physical exam finding that precludes participation, as per investigator
16. Current treatment with CYP2C9 substrates

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2021-06-08 (Actual); Primary Completion 2021-12-16 (Actual); Study Completion 2022-01-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Kaseb, MD, Study Director — Novatek Pharmaceuticals
Locations (3):
- United States (3):
  - Respire Research, San Diego, California
  - L & A Morales Healthcare, Hialeah, Florida
  - United Memorial Medical Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: CSR
Time Frame: November - December 2021

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Active Drug | Placebo
Started | 29 | 26
Completed | 29 | 26
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All patients enrolled, regardless of whether or not they received the assigned treatment
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Drug | Placebo | Total
Number analyzed (Participants) | 29 | 26 | 55
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.48 (19.29) | 45.92 (15.27) | 45.69 (17.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 15 | 31
  Male | 13 | 11 | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 25 | 20 | 45
  Not Hispanic or Latino | 4 | 6 | 10
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 5 | 7
  White | 13 | 12 | 25
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 13 | 9 | 22
Baseline Viral Load assessment [Mean (Standard Deviation); unit: Copies per mililiter of blood] | 16499 (10712) | 15418 (11465) | 16002 (10964)

OUTCOME MEASURES:

1. Primary Outcome: Median Time to Sustained Clinical Response
Description: Measurement of the difference in median time to sustained clinical response in participants taking 3 g TQ Formula (500 mg per capsule, 3 capsules BID) versus participants taking placebo. Sustained clinical response is defined as a reduction of scores to </= 2 on all symptoms of the Modified FLU-PRO Plus.
Time Frame: 21 Days
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Active Drug | Placebo
Number analyzed (Participants) | 29 | 26
Days | 6 [4 to 14] | 8 [5 to 11]

2. Primary Outcome: Number and Percentage of Participants With Overall Adverse Events, Related Adverse Reactions, and Hospitalizations
Description: Number of overall adverse events, related adverse reactions, and hospitalizations reported in participants taking 3 g TQ Formula (500 mg per capsule, 3 capsules BID) versus participants taking placebo. All AEs/SAEs will be captured throughout the study as per schedule of assessments.
Time Frame: From the date of randomization up to Last Visit date on Day-45
Population: This analysis population includes all patients enrolled, randomized, and received at least one dose of the assigned treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Active Drug | Placebo
Number analyzed (Participants) | 29 | 26
Participants | 4 | 7

3. Secondary Outcome: Change of Quantitative Viral Load From Baseline Assessment to Day-14 (Day-14 Minus Baseline)
Description: Measurement of change in quantitative viral load from baseline to Day 14 using RT-PCR (day-14 minus baseline) in participants taking 3 g TQ Formula (500 mg per capsule, 3 capsules BID) versus participants taking placebo with COVID-19 infection.
Time Frame: 14 Days
Measure: Mean (Standard Error); unit: copies/mL
Arm/Group | Active Drug | Placebo
Number analyzed (Participants) | 26 | 23
copies/mL | 13681.67 (13169.47) | 9023.63 (15350.44)

4. Secondary Outcome: Number and Percentages of Study Participants With Viral Clearance
Description: Percentage of negative/undetectable RT-PCR (i.e., viral clearance) on Day-14 in participants taking 3 g TQ Formula (500 mg per capsule, 3 capsules BID) versus participants taking placebo
Time Frame: 14 Days
Population: Patients who had RT-PCR test on Day-14 that was not indeterminate
Measure: Count of Participants; unit: Participants
Arm/Group | Active Drug | Placebo
Number analyzed (Participants) | 21 | 19
Participants | 16 | 11

5. Secondary Outcome: Severity and Change in Covid Symptoms
Description: Measurement of severity of, and change in, Covid-19 symptoms per total score as well as sub-scores (Nose, Throat, Eyes, Chest/Respiratory, Gastrointestinal, Body/Systemic, Taste/Smell) measured through Modified FLU-PRO Plus from Day 1 through Day 14 in participants with COVID-19 infection treated either with 3 g TQ Formula (500 mg per capsule, 3 capsules BID) or placebo.
  1. Total Symptom Score is based on 24 questions with a possible range 0-96
  2. Nose Symptom Score is based on a single question with a possible scale 0-4
  3. Throat Throat Symptom is based on 2 questions with a possible scale 0-8
  4. Respiratory Symptom is based on 7 questions with a possible scale 0-28
  5. GI symptom score is based on 4 questions with a possible scale 0-16
  6. Body/Systemic Symptom Score is based on 8 questions with a possible scale 0-32
  7. Smell/Taste Symptom Score is based on 2 questions with a possible scale 0-8 In each of these scales, higher scores mean higher symptom burden.
Time Frame: 14 Days
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Active Drug | Placebo
Number analyzed (Participants) | 29 | 26
Score on a scale
  Total Symptom Burden within the first 14 days based on 24 questions on a possible scale of 0 to 96 | 12.65 (8.78) | 17.05 (8.78)
  Nose Symptom Burden within the first 14 days based on 1 question on a possible scale of 0 to 4 | 0.54 (0.55) | 0.77 (0.55)
  Throat Symptom Burden within the first 14 days based on 2 questions on a possible scale of 0 to 8 | 0.42 (0.52) | 1.03 (1.55)
  Respiratory Symptom Burden in the first 14 days based on 7 questions on a possible scale of 0 to 28 | 3.48 (4.26) | 4.65 (4.78)
  GI Symptom Burden within the first 14 days based on 4 questions on a possible scale of 0 to 16 | 0.91 (1.10) | 1.48 (1.72)
  Body/systemic Sympt. Burden in the first 14 days based on 8 questions on a possible scale of 0 to 32 | 6.10 (4.34) | 7.08 (5.18)
  Smell/Taste Sympt. Burden in the first 14 days based on 2 questions on a possible scale of 0 to 8 | 1.19 (1.47) | 2.03 (2.09)

6. Secondary Outcome: Correlation Between Covid Symptoms and Viral Load
Description: Correlation Coefficient of quantitative viral load and symptom severity at baseline, at Day 7, and Day 14 in participants taking 3 g TQ Formula (500 mg per capsule, 3 capsules BID) versus participants taking placebo
Time Frame: 14 Days
Measure: Mean (95% Confidence Interval); unit: Correlation Coefficient
Arm/Group | Active Drug | Placebo
Number analyzed (Participants) | 29 | 26
Correlation Coefficient
  Baseline | -0.29 [-0.61 to 0.12] | -0.51 [-0.78 to -0.08]
  Day-7 | -0.51 [-0.77 to -0.12] | -0.53 [-0.80 to -0.09]
  Day-14 | -0.17 [-0.57 to 0.29] | -0.37 [-0.72 to 0.13]

ADVERSE EVENTS:
Time Frame: From the date of Randomization up to the last visit date on Day-45
Description: The trial used CTCAE V5.0
Arm/Group | Active Drug | Placebo
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/29 | 1/26
Other Adverse Events (participants affected / at risk) | 4/29 | 6/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Drug (N=29) | Placebo (N=26)
Hypoxic Respiratory Failure Secondary to COVID Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Drug (N=29) | Placebo (N=26)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Cough after medication. Led to chest pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Sharp chest pain (General disorders) | 1 (1) | 0 (0)
Submandibular abscess (Infections and infestations) | 1 (1) | 0 (0)
couhing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
diarrhea (Gastrointestinal disorders) | 1 (1) | 2 (2)
dry or hacking cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
sleeping more than usual (Nervous system disorders) | 0 (0) | 1 (1)
upper back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
weak (General disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor will be responsible for developing publication procedures and resolving authorship issues. Please refer to your specific contract, grant, and/or Clinical Trials Agreements.

DOCUMENTS (2):
  • Study Protocol (2021-03-25): https://cdn.clinicaltrials.gov/large-docs/77/NCT04914377/Prot_000.pdf
  • Statistical Analysis Plan (2021-09-30): https://cdn.clinicaltrials.gov/large-docs/77/NCT04914377/SAP_001.pdf